CLINICAL TRIAL: NCT02366117
Title: Rehabilitation and Quality of Life in Residential Units for People With Longer Term Mental Health Problems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Direção Geral de Saúde (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 02/2012/CEFCM
Record Dates: First submitted 2015-02-09; First posted 2015-02-19 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Schizophrenia; Mental Disease
Keywords: Quirc; Quality Indiciator in Rehabilitative Care
MeSH Terms: conditions — Schizophrenia; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training (Experimental): Data collected during the first pahse of the study will be presented and discussed in a specialist focus group, which will work with the study team as advisors and trainers, to decide on the type of training to be developed.
  This training intervention will be applied to the facilities presenting half the patient sample size.
  Interventions: Behavioral: Training
- No Training (No Intervention): Facilities representing half the sample size will not be trained as in the Experimental Arm and continue their standard of care for these patients.

INTERVENTIONS:
Behavioral: Training — Adapted training on the patients active participation, rehabilitation, independence, rights and wellbeing.
  Arms: Training

SUMMARY:
The study design is that of a cluster randomised controlled trial

The aims of the study were: 1) to assess the quality of care of the residential units for people with long-term mental disorders; 2) to design a training intervention for the staff of the units in the intervention group; 3) to assess the effectiveness of the intervention 4 and 8 months after it ended.

The main outcome variable was level of activity of the users. Secondary outcome variables were the QuIRC dimensions.

The selection of the sample was by residential units for people with long-term mental disorders.

The inclusion criteria were all the middle and high-support residential units in Portugal. Units that had only one type of service users (e.g., mental retardation, dementia) were excluded.

The quality of care of the units was assessed with the QuIRC filled on line by the managers of the units and validated with Service Users Interview Schedule, a face-to-face interview with the users (users that could not give informed consent or collaborate in the interview were excluded).

DETAILED DESCRIPTION:
The development of community services for treating and rehabilitating people with longer term mental disease, including residential units, is a priority throughout Europe. Recent outcome studies have demonstrated encouraging results in rehabilitation program for most people with schizophrenia, event those with high needs.

Recent legislation in Portugal and the approval of the first Mental Health Plan provided a thrust for developing community services for severe mental patients, specially those directed to patients with schizophrenia or schizoaffective disorders.

The recent National Program for Ongoing Care in Mental Health is a unique opportunity to develop even more residential units and highlights the urgent need to evaluate these facilities.

There are no published studies on the quality of these services, nor the impact that teatment and rehabilitation programs may have on the abilities and negative symptoms of their inpatients because, until recently, their were no reliable instruments for this.

The DEMoB.inc (Development of a European Measure of Best Practice for People with Long Term Mental Illness in Institutional Care) study, a multicentric study financed by the European Comission, between 2007-2010, changed this situation. Its primary goal was the development of a a new instrument for evaluating the quality of the care provided and the quality of life in psychiatric residential units and the social sector. Our team was the portuguese partner for the study.

The final version of the instrument now called QuIRC (Quality Indiciator in Rehabilitative Care) is available in portuguese on www.quirc.com. Several articles on this study have been published.

This set of circumstances opens a unique opportunity:

* The creation of more residential units for longer term mental patients.
* The existence of an instrument designed and developed for assessing these facilities.

The urgent need for assessing the quality of care provided in the facilities and the efectivity of their interventions is the primary goal of this study.

ELIGIBILITY:
Inclusion Criteria:

* Mental Health Problems

Exclusion Criteria:

* Refusal to enter the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of time spent in any activity during a week by patients | Four months
  The percentage of time spent will be measured by the "Time Use Diary" instrument.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Ciências Médicas, Lisbon, Lisbon District, Portugal

REFERENCES:
- [Derived] Cardoso G, Papoila A, Tome G, Killaspy H, King M, Caldas-de-Almeida JM. A cluster randomised controlled trial of a staff-training intervention in residential units for people with long-term mental illness in Portugal: the PromQual trial. Soc Psychiatry Psychiatr Epidemiol. 2017 Nov;52(11):1435-1445. doi: 10.1007/s00127-017-1416-7. Epub 2017 Jun 30. PMID 28667486